CLINICAL TRIAL: NCT07194408
Title: In-Use Tolerance Study Under Dermatological and Pediatric Controls of Sunscreen in Children With Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: RV4620A20230438
Record Dates: First submitted 2025-09-11; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Atopic Dermatitis (AD); SCORAD Index (15-25)
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test group: Children intended to use Sunscreen RV4620A RP2552 product
  Interventions: Other: Sunscreen RV4620A RP2552

INTERVENTIONS:
Other: Sunscreen RV4620A RP2552 — Dermo-cosmetic product, Broadspectrum Sunscreen RV4620A RP2552, very high protection product.
  Instructions for product use given to the subjects: Apply before and during sun exposure, at least twice daily. During sun exposure, applications must be renewed as often as necessary, in particular after swimming, perspiring, towelling, in order to ensure a good protection. On days of bad weather, apply the product in the morning and at the beginning of the afternoon.

SUMMARY:
Atopic dermatitis is a chronic skin condition requiring sun protection, yet research on sunscreen effectiveness and skin tolerance in Atopic Dermatitis is limited. This study evaluates a broad-spectrum SPF50+ sunscreen on 22 children with Atopic Dermatitis, assessing skin tolerance through dermatologic and pediatric controls.

DETAILED DESCRIPTION:
Atopic dermatitis is a chronic skin condition that necessitates sun protection, yet there is limited research on the effectiveness of sunscreens and skin tolerance in Atopic Dermatitis.

Objectives: This study aims to evaluate the tolerance of a broad-spectrum SPF50+ sunscreen in children with Atopic Dermatitis, monitored through dermatological and pediatric assessments.

Methods: This study is conducted on 22 children with Atopic Dermatitis confirmed using the SCORAD index (15-25).

The protocol includes 2 visits and assessments as follow:

* Visit 1: Inclusion (Day 1) - Before and immediately after application (10 to 30 minutes), the investigator conducts a clinical evaluation of the dermatological tolerance of the investigational product. SCORAD evaluation by the dermatologist and pediatrician together is performed on Day 1.
* Home Application Period: Day 1 to Day 22 - Continued application of the sunscreen at home in real conditions of use
* Visit 3: End of Study (Day 22) -The investigators conduct a clinical evaluation of the dermatological tolerance of the investigational product. In addition, a questionnaire is used to evaluate global and perceived efficacy of the sunscreen.

ELIGIBILITY:
Inclusion Criteria:

Criteria related to the population:

* phototype: I to IV;
* face and body skin type: all skin types;
* subjects must be registered with health social security or health social insurance (if required by national regulations);
* subjects' parent(s)/ legal representatives having signed their written Informed Consent form for their participation in the study and a photograph authorization;
* subjects' parent(s)/ legal representatives certifying the truth of the personal information declared to the Investigator;
* Health Status: Considered a "healthy subject" by the Investigators (excluding SCORAD considerations).

Criteria Related to Atopic Dermatitis:

- Subject must present atopic dermatitis according to the U.K Working Party's Diagnostic Criteria for Atopic Dermatitis, with mild atopic dermatitis indicated by a SCORAD score of 15 to 25 (inclusive), determined by a dermatologist and a pediatrician together.

Non-Inclusion Criteria:

Criteria Related to Population:

* Subjects who have participated in another clinical trial within the week before the inclusion visit, or for a longer period if deemed necessary by the Investigator.
* Subjects currently participating or planning to participate in another clinical trial during the study, either in the same or a different investigation center.

Criteria Related to Subject's Health:

* Subjects experiencing a flare of atopic dermatitis.
* Subjects with dermatological conditions that may interfere with study data or are considered hazardous by the Investigator (e.g., pityriasis versicolor, severe pigmentation disorders such as vitiligo, melasma, multiple lentigines, numerous or large congenital nevi).
* Subjects with a personal medical history that may interfere with study data or is incompatible with study requirements (except if required by the Sponsor, e.g., atopic dermatitis).

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be recruited from the investigation centre's panel. They will be selected on the basis of inclusion and non-inclusion criteria specific to the study and on their ability to comply with the constraints required by the protocol. They will be definitely included in the study after a specific interview and a clinical examination.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

PRIMARY OUTCOMES:
Global tolerance assessment by the investigator | At the end of the study, after Last Patient Out, (after Day 22)
  Global tolerance is assessed on the "tolerance population" which includes all the subjects who applied at least once investigational product.
  This assessment allows for attribution of one of the 5 levels : excellent, very good, good, moderate, bad.

SECONDARY OUTCOMES:
Evaluation Global Acceptability of the Sunscreen RV4620A - RP2552 | Visit 3 (Day 22)
  The subjects' parent(s)/ legal representatives give their global appreciation about the product with positive and negative feedback. According to the items, the subjects' parent(s)/ legal representatives have to answer opened questions and a question using a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Insight Research, Quatre Bornes, Mauritius, Mauritius